CLINICAL TRIAL: NCT07106645
Title: Transcranial Magnetic Stimulation in Anorexia Nervosa: A Double-Blind Randomized Study on the Efficacy of Intermittent Theta Burst Stimulation of the Right Parietal Lobe
Brief Title: Intermittent Theta Burst Transcranial Magnetic Stimulation of the Right Parietal Lobe in Anorexia Nervosa
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Padova (Other)
Collaborators: Azienda Ospedaliera di Padova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 6168/EST/25
Record Dates: First submitted 2025-07-18; First posted 2025-08-06 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-07

CONDITIONS: Anorexia Nervosa
Keywords: psychiatry; eating disorders; neurostimulation; TMS; Transcranial Magnetic Stimulation; Anorexia Nervosa
MeSH Terms: conditions — Anorexia Nervosa; Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Each patient will be randomly assigned to one of two conditions: (1) active iTBS; (2) sham stimulation
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Both patients and experimenters will be blind to the condition
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- active iTBS (Experimental): Patients in this condition will undergo 20 sessions of iTBS over the right posterior parietal lobe, one per day for 20 consecutive working days (4 weeks)
  Interventions: Device: Active iTBS
- sham stimulation (Active Comparator): Patients in this condition will undergo 20 sessions of sham stimulation over the right posterior parietal lobe, one per day for 20 consecutive working days (4 weeks)
  Interventions: Device: Sham stimulation

INTERVENTIONS:
Device: Active iTBS — Patients in this condition will undergo 20 sessions of iTBS, one per day for 20 consecutive working days (4 weeks). Each visit will last approximately 20 minutes, including preparation, 3 minutes of stimulation, and debriefing. The coil position will be identified using a neuronavigation system based on each participant's MRI. Intermittent theta burst stimulation will involve the delivery of triplets of pulses at 50 Hz, repeated at 5 Hz, at 100% of the individual motor threshold.
  Arms: active iTBS
Device: Sham stimulation — Patients in this condition will undergo 20 sessions of sham stimulation, one per day for 20 consecutive working days (4 weeks). Each visit will last approximately 20 minutes, including preparation, 3 minutes of stimulation, and debriefing. The coil position will be identified using a neuronavigation system based on each participant's MRI. Sham stimulation will be identical to active stimulation, with the only difference being the use of a sham coil, which produces the same sound as the real coil without generating a magnetic field
  Arms: sham stimulation

SUMMARY:
Anorexia Nervosa is a psychiatric disorder characterized by high rates of chronicity, significant societal costs, and one of the highest mortality rates among psychiatric illnesses. Despite therapeutic advances, treatment outcomes remain poor, with high relapse rates and full recovery achieved in only 50% of cases.

Recent cognitive, behavioral, and neuroimaging studies suggest that Anorexia Nervosa may involve dysfunction in a posterior parietal network responsible for multisensory integration. This network plays a pivotal role in bodily self-representation and the modulation of environment-body interactions, and may therefore be directly implicated in two core symptoms of the disorder: distorted body image representation and dietary restriction. Given these insights, Transcranial Magnetic Stimulation (TMS) - an established neuromodulation technique with proven efficacy in various psychiatric disorders - emerges as a promising investigational intervention. The aim of this study is to evaluate the feasibility and therapeutic efficacy of a protocol of intermittent Theta Burst Stimulation (iTBS) targeting the right posterior parietal lobe in patients with Anorexia Nervosa. The active iTBS protocol will be compared to a sham (placebo) stimulation as a control condition.

DETAILED DESCRIPTION:
Patients with anorexia nervosa will be recruited from the Eating Disorder Unit of Padova Hospital. Inclusion criteria will be: (1) current diagnosis of anorexia nervosa according to DSM-5 criteria; (2) 18 years or older; (3) failure of an outpatient treatment cycle lasting at least 3 months. Exclusion criteria will be: (1) Presence of significant neurological comorbidities or severe/unstable systemic diseases, (2) Diastolic blood pressure <60 mmHg or heart rate <60 bpm, (3) diagnosis of psychosis or substance abuse disorders, (4) history of hypomanic/manic episodes (5) Current suicidal ideation, (6) known contraindications to TMS (epilepsy, head trauma with loss of consciousness, severe/frequent headaches, cochlear implants, pacemakers, pregnancy, metallic implants, implanted neurostimulators)

Each patient will be randomly assigned to one of two conditions: active iTBS or sham stimulation

iTBS protocol: Patients in this condition will undergo 20 sessions of iTBS, one per day for 20 consecutive working days (4 weeks). Each visit will last approximately 20 minutes, including preparation, 3 minutes of stimulation, and debriefing. The coil position will be identified using a neuronavigation system based on each participant's MRI. Intermittent theta burst stimulation will involve the delivery of triplets of pulses at 50 Hz, repeated at 5 Hz, at 100% of the individual motor threshold.

Sham Stimulation: Patients in this condition will undergo the same protocol (20 sessions of TMS), with the only difference being the use of a sham coil, which produces the same sound as the real coil without generating a magnetic field

Patients in both conditions will complete a baseline assessment (Day 0), an end-of-treatment assessment (Week 4), and a follow-up assessment (4 months after the end of treatment).

All the assessments will include:

Clinical interview with a psychiatrist who is blind to the stimulation condition. During the interview, the clinician will also record the patients' weight and height to calculate Body Mass Index (BMI).

Depression Anxiety Stress Scales - 21 items (DASS-21): a validated 21-item scale for assessing depression, anxiety, and stress.

Eating Disorders Inventory (EDI-I): a validated 64-item scale for assessing eating disorder psychopathology.

Body Attitude Questionnaire: a validated questionnaire on body dissatisfaction and body perception.

Wisconsin Card Sorting Task (WCST): assessment of set-shifting abilities.

Rey-Osterrieth Complex Figure Test: assessment of central coherence.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria will be: (1) current diagnosis of anorexia nervosa according to DSM-5 criteria; (2) 18 years or older; (3) failure of an outpatient treatment cycle lasting at least 3 months

Exclusion Criteria:

* Exclusion criteria will be: (1) Presence of significant neurological comorbidities or severe/unstable systemic diseases, (2) Diastolic blood pressure <60 mmHg or heart rate <60 bpm, (3) diagnosis of psychosis or substance abuse disorders, (4) history of hypomanic/manic episodes (5) Current suicidal ideation, (6) known contraindications to TMS (epilepsy, head trauma with loss of consciousness, severe/frequent headaches, cochlear implants, pacemakers, pregnancy, metallic implants, implanted neurostimulators)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2027-01-15 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Body Mass Index (BMI) | Day 0 (baseline), Week 4 (end of treatment), Week 20 (4-month follow-up)
  BMI will be calculated from patients' height and weight using the formula: weight (kg) divided by height (m) squared.

SECONDARY OUTCOMES:
Change from baseline in depression, anxiety and stress | Day 0 (baseline), Week 4 (end of treatment), Week 20 (4-month follow-up)
  The DASS-21 is a validated self-report instrument consisting of three subscales assessing symptoms of depression, anxiety, and stress. The score of each subscale can range from 0 to 42, with higher scores representing higher levels of psychopathology.
Change from baseline in eating disorder psychopathology | Day 0 (baseline), Week 4 (end of treatment), Week 20 (4-month follow-up)
  The EDI-I is a 64-item self-report scale for the assessment of eating disorder psychopathology. The scale comprises 8 subscales (drive for thinness, bulimia, body dissatisfaction, ineffectiveness, perfectionism, interpersonal distrust, interoceptive awareness, maturity fears). Total score ranges from 64 to 384 and greater scores indicate greater psychopathology
Change from baseline in body dissatisfaction and perception | Day 0 (baseline), Week 4 (end of treatment), Week 20 (4-month follow-up)
  The Body Attitude Questionnaire is a 26 item self-report scale for the assessment of body dissatisfaction and perception. The questionnaire comprises 3 subscales (body satisfaction, body concern, body distortion). Total score ranges from 26 to 130 and higher scores indicate greater body dissatisfaction and concern.
Change from baseline in cognitive flexibility | Day 0 (baseline), Week 4 (end of treatment), Week 20 (4-month follow-up)
  The Wisconsin Card Sorting Task is a well-validated neuropsychological task for the assessment of cognitive flexibility. As outcome variables, the number of perseverative responses and perseverative errors will be taken into account.
Change from baseline in central coherence | Day 0 (baseline), Week 4 (end of treatment), Week 20 (4-month follow-up)
  The Rey-Osterrieth complex figure is a well-validated neuropsychological test for the assessment of visuospatial functioning and memory. As outcome variables, the indexes of central coherence in both the copy and memory phase will be taken into account.

OTHER OUTCOMES:
feasibility and acceptability of iTBS treatment | 4 weeks
  percentage of patients who will complete the intervention

CONTACTS AND LOCATIONS:
Overall Officials: Enrico Collantoni, MD, PhD, Principal Investigator — University of Padova
Locations (1):
- Psychiatric Unit, Padua, Padova, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Meregalli V, Gentili S, Menardi A, Vallesi A, Olivo D, Manara R, Serino A, Risso G, Sambataro F, Favaro A, Collantoni E. Individualized targeting of the posterior parietal cortex with intermittent theta burst stimulation in anorexia nervosa: a randomized, double-blind, sham-controlled protocol. Front Neurosci. 2026 Jan 21;19:1733280. doi: 10.3389/fnins.2025.1733280. eCollection 2025. PMID 41648851